CLINICAL TRIAL: NCT03566030
Title: Real-life Data of Switching From Tenofovir Disoproxi Fumarate (TDF) to Tenofovir Alafenamide (TAF) in Virologically Suppressed Chronic Hepatitis B Patients With Antiviral Resistance
Brief Title: Switching From Tenofovir Disoproxi Fumarate to Tenofovir Alafenamide in Chronic Hepatitis B Patients With Antiviral Resistance
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-320-4406
Record Dates: First submitted 2018-05-22; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B; Antiviral Drug Adverse Reaction
Keywords: Hepatitis B; Tenofovir Disoproxil Fumarate; Tenofovir Alafenamide; Switch
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tenofovir Disoproxil Fumarate 300 mg QD: Administered Tenofovir Disoproxil Fumarate 300 mg QD
  Interventions: Drug: Tenofovir disoproxil fumarate 300mg
- Tenofovir Alafenamide: Administered Tenofovir Alafenamide 25 mg QD
  Interventions: Drug: Tenofovir Alafenamide 25 mg

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate 300mg — Administered Tenofovir disoproxil fumarate 300 mg QD
  Other Names: TDF
  Groups: Tenofovir Disoproxil Fumarate 300 mg QD
Drug: Tenofovir Alafenamide 25 mg — Administered Tenofovir Alafenamide 25 mg QD
  Other Names: TAF
  Groups: Tenofovir Alafenamide

SUMMARY:
* To evaluate the efficacy of switching to tenofovir alafenamide (TAF) 25 mg QD versus continued tenofovir disoproxil fumarate (TDF) 300 mg QD in CHB patients with antiviral resistance, as determined by the proportion of virologically suppressed patients at week 48
* To evaluate the safety and tolerability of switching to TAF 25 mg QD versus continuing TDF 300 mg QD in antiviral-resistant subjects with chronic HBV at week 48

DETAILED DESCRIPTION:
The investigators will conduct a multicenter observational study to evaluate the safety and efficacy of TAF 25 mg QD in chronic hepatitis B patients with antiviral resistance who switch from TDF to TAF. The safety and antiviral activity will be assessed as a part of routine medical care. Subjects will be obtained from an existing cohort of patients treated with a TDF-based regimen due to antiviral resistance, which has been supported by Gilead (IN-US-174-1255).

It is anticipated that approximately 300 CHB patients with antiviral resistance taking TDF 300 mg QD will be enrolled in this study. All consecutive patients will be allocated to receive either TAF 25 mg QD or TDF 300 mg QD (possibly 50% vs. 50%, the proportion of patients enrolled in the study is an estimate based on the clinical experience.), according to the decision of the individual patients and their physicians, with informed consent. Patients are switched independently based on physicians discretion/decision prior to study enrollment, and the study protocol would NOT have any influence over the process.

All consecutive patients will be prospectively monitored every 6 months during the first year and thereafter every 6 months up to 3 years. At each visit, a routine examination and determination of biochemical and virological parameters (HBV DNA level, HBeAg, anti-HBe, HBsAg [quantitatively, if available], and anti-HBs) will be performed. Lab tests and markers will be routinely monitored every 6 months.

Recruitment method: In this study, we plan to use an existing cohort of patients treated with a TDF-based regimen due to antiviral resistance (IN-US-174-1255). Data on all consecutive patients currently receiving TDF due to antiviral resistance at enrollment will be followed up prospectively every 3-6 months for 2 years. The patients will be recruited consecutively. Patients will be recruited only after the treatment decision has been made. No aspect of this study will interfere with or influence routine medical practice.

Number of study sites: At least seven representative institutes in South Korea. Target population: Korean adult subjects with CHB receiving TDF due to antiviral resistance.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
* Adult male and non-pregnant, non-lactating female subjects, ≥20 years of age based on the date of the screening visit.
* Documented evidence of chronic HBV infection previously
* TDF monotherapy, TDF-based combination therapy, or switching to TAF at least 4 weeks prior to screening in virologically suppressed chronic hepatitis B patients with multi-antiviral resistance
* Must be willing and able to comply with all study requirements

Exclusion Criteria:

• Co-infection with HCV, HDV, HIV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will conduct a multicenter observational study to evaluate the safety and efficacy of TAF 25 mg QD in chronic hepatitis B patients with antiviral resistance who switch from TDF to TAF. Subjects will be obtained from an existing cohort of patients treated with a TDF-based regimen due to antiviral resistance, which has been supported by Gilead (IN-US-174-1255).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Serum HBV DNA level | at week 48
  The proportion of subjects who achieve a sustained serum HBV DNA level < 20 IU/mL (undetectable serum HBV DNA by PCR)

SECONDARY OUTCOMES:
Serum HBV DNA level | at week 96
  The proportion of subjects who achieve a sustained serum HBV DNA level < 20 IU/mL (undetectable serum HBV DNA by PCR)
Hip and spine BMD | at 48, 96 week
  The percent change in hip and spine BMD from baseline
Serum eGFR | at 24, 48, 72, and 96 week
  The change in serum eGFR (Cockcroft-Gault method) from baseline
Serum creatinine & PO4 level | at 24, 48, 72, and 96 week
  The change in serum creatinine & PO4 from baseline